CLINICAL TRIAL: NCT06861673
Title: COnCOmitaNt Pulse Field Ablation Based pUlmonary Vein Isolation and lefT Atrial Appendage Closure - The COCONUT Study
Brief Title: COCONUT Study Concomitant PVI and LAAC
Acronym: COCONUT
Status: Recruiting | Type: Observational
Sponsor: Asklepios proresearch (Industry)
Responsible Party: Principal Investigator, Prof. Christian-Hendrik Heeger, Prof. Dr., Asklepios proresearch
Other Study IDs: COCONUT register
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Concomitant PVI plus LAAC
  Interventions: Device: Pulmonary vein isolation

INTERVENTIONS:
Device: Pulmonary vein isolation — concomitant PVI and LAAC

SUMMARY:
In patients with non-valvular AF, at high stroke risk, and who are ineligible for long-term oral anticoagulation LAAC could be an alternative to anticoagulation and safety and efficacy has been shown in several studies and registries.8 While PVI and LAAC are both conducted in the left atrium and share the same access route, a combined concomitant approach might be beneficial for patients but is not conventionally practiced. Due to significantly shorter procedures times and high safety profile PFA based catheter ablation may be advantageous for the combined approach of PVI and LAAC. We are performing a word-wide, retrospective, multicenter registry study focusing on patients with concomitant Farapulse PFA based PVI and LAAC (WATCHMAN Flx, Boston Scientific). To evaluate safety, efficacy and efficiency in a multicenter study the COCONUT study was conducted.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) ablation by pulmonary vein isolation and left atrial appendage closure (LAAC) are increasingly performed as individual procedures. However, there are several studies which investigated a combined concomitant approach of perfoming a cryoballoon or radiofrequency based PVI and an interventional LAAC in one procedure and safety and efficacy has been shown. 1,2,3,4 The novel ablation modality pulsed field ablation (PFA) has significantly reduced procedure duration and potentially increased safety due a specific ablation of cardiac tissue with sparing smooth muscle cells and nervous cells.6 With currently >100.000 treated patients most experience is currently available for the Farapulse PFA system (Boston Scientific). The MANIFEST-PF and MANIFEST 17K registries showed an excellent safety and efficacy profile of this novel ablation technology.6,7 In patients with non-valvular AF, at high stroke risk, and who are ineligible for long-term oral anticoagulation LAAC could be an alternative to anticoagulation and safety and efficacy has been shown in several studies and registries.8 While PVI and LAAC are both conducted in the left atrium and share the same access route, a combined concomitant approach might be beneficial for patients but is not conventionally practiced. Due to significantly shorter procedures times and high safety profile PFA based catheter ablation may be advantageous for the combined approach of PVI and LAAC. We are performing a word-wide, retrospective, multicenter registry study focusing on patients with concomitant Farapulse PFA based PVI and LAAC (WATCHMAN Flx, Boston Scientific). To evaluate safety, efficacy and efficiency in a multicenter study the CONOCNUT study was conducted. Two months after successful PVI and LAAC the OAC therapy could be terminated which might be beneficial for the patients especially for those with a higher bleeding risk. Further potential benefits are the reduction of periprocedural complications. Furthermore, economic factors could be beneficial due to only one concomitant procedure with one hospital stay instead of two procedures with two hospital stays.

ELIGIBILITY:
Inclusion Criteria:

Indicatio for PVI and LAAC

Exclusion Criteria:

Not eligible for any of the procedures PVI and LAAC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with AF and PVI plus LAAC
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety | within 3 days
  Peri- and postprocedural complications:
  Rate of: pericardial tamponade, pericardial effusion, Venouse access site haematoma
Efficacy | one year
  Sinus rhythm after one year

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepios Klinik Altona, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No